CLINICAL TRIAL: NCT02767284
Title: UCST Studie 1 - Jämförande Studie Mellan några Befintliga Och Nyutvecklade Metoder för Att mäta Den Spektrala kontrastkänslighetsfunktionen Hos människa
Brief Title: A Comparative Study of Six Methods to Measure Human Contrast Vision
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: UCST-01.2014
Record Dates: First submitted 2016-05-04; First posted 2016-05-10 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Methods to Measure Contrast Vision
Keywords: Contrast Sensitivity; Diagnostic Techniques, Ophthalmological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- UCST-V1 (Experimental): The UCST-V1 contrast sensitivity test, used to measure CSF thrice in each eye at two occasions in every treatment sequence (multi-period crossover)
  Interventions: Device: UCST-V1
- UCST-V2 (Experimental): The UCST-V2 contrast sensitivity test, used to measure CSF thrice in each eye at two occasions in every treatment sequence (multi-period crossover)
  Interventions: Device: UCST-V2
- UCST-V3 (Experimental): The UCST-V3 contrast sensitivity test, used to measure CSF thrice in each eye at two occasions in every treatment sequence (multi-period crossover)
  Interventions: Device: UCST-V3
- Quick-CSF (Experimental): The Quick-CSF test, used to measure CSF thrice in each eye at two occasions in every treatment sequence (multi-period crossover)
  Interventions: Device: Quick-CSF (QCSF)
- Pelli-Robson (Active Comparator): The Pelli-Robson contrast sensitivity test, used to measure CSF thrice in each eye at two occasions in every treatment sequence (multi-period crossover)
  Interventions: Device: Pelli-Robson
- Optec 6500 (Active Comparator): The Optec 6500 contrast sensitivity test, used to measure CSF thrice in each eye at two occasions in every treatment sequence (multi-period crossover)
  Interventions: Device: Optec 6500

INTERVENTIONS:
Device: UCST-V1 — A previously developed device, Uppsala Contrast Sensitivity Tester - UCST-V1, that quickly measures the human CSF in one stimulus.
  Arms: UCST-V1
Device: UCST-V2 — A refined version of the UCST-V1 that randomizes frequency order.
  Arms: UCST-V2
Device: UCST-V3 — A version that utilises eye-tracking technology to make the measurements more accurate.
  Arms: UCST-V3
Device: Quick-CSF (QCSF) — A fast contrast sensitivity measurement method using a Bayesian algorithm.
  Arms: Quick-CSF
Device: Pelli-Robson — A standard method developed using a Sloan-letter chart with decreasing contrast.
  Arms: Pelli-Robson
Device: Optec 6500 — A standard test using sinusoidal gratings to measure the contrast sensitivity function.
  Arms: Optec 6500

SUMMARY:
This study evaluates the relative performance of different methods to measure the human spectral contrast sensitivity function (CSF).

DETAILED DESCRIPTION:
The human spectral contrast sensitivity function (CSF) is a better way to estimate human vision than letter charts commonly used by ophthalmologists, optometrists and opticians.

The current methods used to measure the CSF are often unreliable, due to high variability between measurements. This study will compare four (4) new tests with two (2) currently used standard tests. The contrast sensitivity function will be measured using all of the six (6) methods three times (3) in each of the two (2) eyes at two (2) occasions. Each subjects CSF will be measured 6x3x2x2 = 72 times.

In addition, for each of the CSF measurements, the time used to measure the CSF and number of background variables for the subjects will be recorded.

After informed consent is obtained, the subjects will undergo a visual examination. If they match the inclusion criteria they will be included. At that time or at their earliest possible convenience, their CSF will be measured using the six methods and some background information will be recorded.

The follow-up measurement occasion will occur between 4 to 6 weeks (28 to 42 days) after the first.

To facilitate comparison with previous studies, the CSF-measurements (in rel. contrast/cycles/degree) will be converted to a log (Base 10 logarithm) scale. The unit will thus be log CSF (LCSF) [log[relative contrast]/log[cycles/per degree]].

ELIGIBILITY:
Inclusion Criteria:

* Normal best corrected visual acuity: LogMAR = 0
* No current or previous eye disease in either eye.
* Student at Uppsala University

Exclusion Criteria:

* Previous surgery in any eye
* Inability to follow the test procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Average time (in seconds) used to measure the contrast sensitivity function for one eye for each method | At end of data collection (up to 12 months after first subject is included)
Average area under the curve for the log contrast sensitivity function (AULCSF) in one eye for each method | At end of data collection (up to 12 months after first subject is included)
  The area-under-curve of the LCSF, calculated from the measured CSF.

SECONDARY OUTCOMES:
Sources of variability of the average time used to measure the contrast sensitivity function [seconds squared] | At end of data collection (up to 12 months after first subject is included)
  The factors occasion, eye, acuity, measurement order, sex,examiner will used in an ANOVA
Sources of variability of the average area under the curve for the log contrast sensitivity function [AULCSF squared] | At end of data collection (up to 12 months after first subject is included)
  The factors occasion, eye, acuity, measurement order, sex,examiner will used in an ANOVA

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Per Söderberg, M.D PhD, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Anonymous or pseudo-anonymous data will be available on request or in a repository.